CLINICAL TRIAL: NCT01738126
Title: fMRI and DTI of Cerebellar Responses to Pain in the Human Trigeminal System
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Eric Alan Moulton, Assistant Professor, Mclean Hospital
Other Study IDs: NIH-K01DA025289
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Cerebellum and Pain in Healthy Volunteers.
Keywords: cerebellum; fMRI; DTI; pain; heat; noxious; aversion; unpleasantness; anger; aversive stimulus; motor; human; image analysis; perception; central nervous system; sensory; somatosensory cortex; trigeminal system; white matter
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
This K01 application is designed to prepare the applicant with the skills necessary to establish an independent research program on pain--related processing in the cerebellum. Although pain studies using functional imaging in humans consistently find cerebellar activation, the role of this structure during pain is unknown. In such studies, speculation regarding the cerebellum's function during a painful event is often influenced by its reputation as a coordinator of motor function, though animal studies have indicated that it may also modulate the neural encoding of noxious stimuli. The candidate has published work that indicates a functional dichotomy in the way the cerebellum responds to experimental pain in healthy subjects and neuropathic pain patients. This suggests that the cerebellum has been overlooked as a potential pain processing area, and research into this area could lend invaluable insight into the basic physiological circuitry involved with pain and its modulation.

The hypothesis of this project is that the cerebellum serves as an integrator of aversive stimuli and adaptive motor behavior, and may modulate the emotional and cognitive experience that distinguishes the perception of pain from the appreciation of innocuous sensory stimulation. A human trigeminal model of experimental pain will be used, as all the pain---related circuitry involved can be imaged along with the cerebellum at the same time. The specific aims are (1) to map cerebellar activations related to sensory coding of noxious stimuli and to correlate functional activity with anatomical connectivity using functional magnetic resonance imaging (fMRI) and diffusion tensor imaging (DTI); (2) to distinguish between pain and its anticipation based on cerebellar responses and connectivity; and (3) to determine whether physical pain and aversive images engage similar circuitry in the cerebellum. To accomplish these aims, the candidate will need to expand his background in fMRI of cortical and brainstem pain processing to encompass cerebellar physiology, become proficient in DTI analysis, and learn the white matter connectivity to and from the cerebellum. The research environment at McLean Hospital and the other affiliates of the Harvard Medical School system will provide the candidate with the resources to reach his aims within 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed subjects
* Good physical health
* No history of claustrophobia
* English speaking and reading ability sufficient to comprehend consent without assistance

Exclusion Criteria:

* History of drug abuse or positive drug screen
* Magnetic Implants of any type (including dental bridges, crowns, retainers, orthodontic devices, etc)
* Weight > 285 pounds (weight limit of the fMRI table)
* Positive pregnancy screen
* Beck Depression Inventory II (BDI-II) score > 25 (moderate to severe depression)
* History of primary depression, anxiety disorders, or mood disorders
* Prolonged use of antidepressants or anticonvulsants
* Evidence of local pathology; e.g. cancer affecting the face
* History of systemic disorders, e.g. multiple sclerosis
* History of chronic pain, e.g. back pain
* History of primary headache, e.g. migraine, tension-type headache
* Recent orofacial surgery or trauma
* History of central origin disorders, eg. stroke
* History of dermatological hypersensitivity in the facial area
* History of Eczema
* Significant medical history of seizure disorder, diabetes, cardiac disease including coronary artery disease, psychiatric problems; respiratory problems, liver disease, etc.
* Significant alcohol history (ingestion of 5 or more glasses (>40 oz) of alcohol per week)
* Claustrophobia
* Pregnancy
* Smokers
* Tattoos containing metallic ink on the neck, shoulders, upper arm and head (which could become heated up in the scanner, and potentially cause blistering or burning)
* Cardiac pacemakers
* Aneurysm clips and other vascular stents, filters, clips or other devices
* Prosthetic heart valves
* Other prostheses
* Neuro-stimulator devices
* Implanted infusion pumps
* Cochlear (ear) implants
* Ocular (eye) implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* Repeated monthly usage of the ovulation test kit fails to detect a luteinizing hormone surge (for females not on contraception only)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy human volunteers
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-05; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Whole brain functional magnetic resonance imaging (fMRI) data | 1 year
  fMRI data is used to indirectly measure neurophysiological responses in the brain using the blood oxygen level dependent (BOLD) signal.
Pain ratings | 1 year
  Subjective pain ratings elicited by experimental stimuli.
Whole-brain diffusion tensor imaging (DTI) data | 1 year
  DTI data measures the integrity of white matter tracts in the brain, based on principles of water diffusion.